CLINICAL TRIAL: NCT05109169
Title: Multimodal METformin and FINGER Lifestyle Intervention to Prevent Cognitive Impairment and Disability in Older Adults at Risk for Dementia: a Phase IIb Multi-national Randomised, Controlled Trial
Brief Title: METformin and FINGER Intervention to Prevent Cognitive Impairment and Disability in Older Adults at Risk for Dementia
Acronym: MET-FINGER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Alzheimer's Association (Other); Alzheimer's Drug Discovery Foundation (Other); Alzheimerfonden (Unknown); Region Stockholm (Other Government); Merck KGaA, Darmstadt, Germany (Industry); Finnish Institute for Health and Welfare (Other Government); Fingers Brain Health Institute (Other); Karolinska University Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21CX6667; 2021-005213-14 (EudraCT Number); 2022-500438-27-01 (Other: EMA (EU-CT number))
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Decline; Cognitive Impairment; Dementia
Keywords: Dementia prevention; FINGER multidomain lifestyle intervention; Metformin; World-Wide FINGERs; Drug repurposing
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: Participants are initially randomized 1:1 to two parallel arms:
  * self-guided multidomain lifestyle intervention
  * FINGER 2.0 multidomain lifestyle-based intervention
  Participants in the FINGER 2.0 intervention who are eligible for metformin treatment will be further randomized 1:1:1 to either:
  * metformin 2000mg/day
  * metformin 1000mg/day
  * placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Lifestyle intervention: participants will not be told to what intervention group they have been assigned and outcome assessors will be blinded to the lifestyle intervention group allocation.
  Metformin/placebo treatment within the FINGER 2.0 intervention group: double blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-guided multidomain lifestyle intervention (Sham Comparator): In this group, participants will build their own healthy lifestyle program based on standard healthy lifestyle advice that they will receive at individual consultations with the study physician/nurse as part of the study visits, covering four main components (diet, physical activity, cognitive training, and cardiovascular/metabolic risk monitoring). The intervention duration is 2 years.
  Interventions: Other: Self-guided multidomain lifestyle intervention
- FINGER 2.0 multidomain lifestyle-based intervention (Active Comparator): Within this group, participants will receive a structured intensive lifestyle intervention through individual consultations and group meeting sessions. Four main lifestyle components will be included (diet, physical activity, cognitive training, and cardiovascular/metabolic risk monitoring) as well as social interaction through the group meetings/sessions.
  In this group, participants eligible for metformin treatment will be further randomised to either:
  * 2000mg/day
  * 1000mg/day
  * placebo.
  Metformin and placebo will be dispensed every 3 months, both administered orally. The intervention duration is 2 years
  Interventions: Combination Product: FINGER 2.0 multidomain lifestyle-based intervention

INTERVENTIONS:
Combination Product: FINGER 2.0 multidomain lifestyle-based intervention — Multimodal lifestyle-based precision prevention intervention, including:
  * Optimized FINGER multidomain lifestyle intervention (diet, physical activity, cognitive training and cardiovascular/metabolic risk monitoring and social interaction)
  * Metformin (Glucophage® XR)
  Arms: FINGER 2.0 multidomain lifestyle-based intervention
Other: Self-guided multidomain lifestyle intervention — Participants build their own healthy lifestyle program based on standard healthy lifestyle advice on diet, physical activity, cognitive training and cardiovascular/metabolic risk
  Arms: Self-guided multidomain lifestyle intervention

SUMMARY:
Dementia is the main cause of disability in older adults, currently affecting about 50 million people world-wide with this number estimated to triple in the next 30 years. In MET-FINGER, we aim to understand whether the FINGER 2.0 multidomain intervention, combining healthy lifestyle changes and a drug for diabetes (metformin), may help reduce the risk of dementia and improve health and independence among older adults.

The study primary objective is to test the effect of the intervention, compared to healthy lifestyle advice, on the change in cognition, measured as a composite score including 14 of neuropsychological/cognitive tests. The secondary objective is to test the intervention effect on change in individual cognitive domains, functioning level, and risk factors for dementia (e.g., lifestyle, medical, and psychosocial). To this aim, a range of personal/health-related data and blood samples, will be collected. Potential interactions between metformin and lifestyle changes; potential disease-modifying effects; and feasibility of the metformin + lifestyle combination will be explored.

600 older people with risk factors for dementia, but without dementia/substantial cognitive impairment, will be recruited in the United Kingdom, Finland, and Sweden (at least 50% with higher genetic risk of Alzheimer's Disease/dementia based on the Apolipoprotein E (APOE) gene). Participants will be randomly assigned 1:1 to either a self-guided multidomain lifestyle intervention or to the FINGER 2.0 multidomain lifestyle-based intervention. Outcome assessors will be blinded to group allocation. Within the FINGER 2.0 intervention group, participants at increased risk of diabetes, will be randomly assigned 1:1:1 to either the metformin 2000mg/day, metformin 1000mg/day, or placebo group (double blinded). The intervention duration is 24 months.

The lifestyle intervention includes four main components: physical exercise, diet, brain training and health checks. In the self-guided group, participants will create their own program, based on health advice and recommendations which will be provided during the study. In the FINGER 2.0 intervention group, participants will receive intensive lifestyle guidance, and participate in structured activities, which will be as tailored as possible on each person's daily habits and needs.

Over the 2-year study period, all participants will attend four assessment visits: baseline, 6-, 12-, and 24-months.

DETAILED DESCRIPTION:
After being identified and pre-screened in relevant registers, potential participants will undergo a screening assessment (after providing informed consent for the screening procedures) where inclusion criteria related to both cognition and cardiovascular/lifestyle risk factors will be checked. Participants meeting the inclusion criteria will undergo the exclusion criteria assessment with the study physician.

Eligible participants will be invited to the baseline visit where informed consent for the full study will be signed, baseline assessment will be conducted, and participants will be randomized to either the FINGER 2.0 multidomain lifestyle-based intervention or self-guided multidomain lifestyle intervention group. Based on the results of the baseline assessment, the eligibility to the metformin/placebo treatment will be assessed in all participants randomized to the FINGER 2.0 intervention group. Eligible participants will be further randomized to one of the three metformin treatment groups (metformin 2000mg/day, metformin 1000mg/day, or placebo). Non eligible participants will continue the study by following the structured lifestyle intervention alone.

In the self-guided intervention group, participants will build their own healthy lifestyle program based on standard healthy lifestyle advice that they will receive at individual consultations with the study physician/nurse as part of the visits.

Within the FINGER 2.0 intervention group, participants will be invited to attend individual consultations and group meeting sessions in relation to the four intervention components (diet, physical activity, cognitive training, and cardiovascular/metabolic risk monitoring). As part of the physical activity component, group training sessions with a physiotherapist/professional trainer will be organized both at a gym as well as online. Within the cognitive training component, participants will have access to an online cognitive training program for independent training sessions. Individually tailored recommendations and plans will be provided to each participant.

Metformin and placebo will be dispensed every 3 months, both administered orally. The active drug is Glucophage® XR 500. All participants randomized to the metformin/placebo groups will receive 4 identical tablets per day as follows:

* 2000mg/day: 4x500mg metformin
* 1000mg/day: 2x500mg metformin + 2x500mg placebo
* Placebo: 4x500mg placebo.

Metformin will be titrated weekly from 500mg/day up to 2000mg/day over 4 weeks. Participants who do not tolerate the treatment will be allowed to remain in the study either in a lower dose treatment group, or receiving the structured lifestyle intervention only.

Participants will not be actively told to what lifestyle intervention group they have been assigned and assessors for primary and secondary outcomes will be blinded to the lifestyle group allocation. The metformin/placebo treatment will be conducted in double blind.

ELIGIBILITY:
Inclusion Criteria:

* Main inclusion criteria (all participants)

  1. Age 60-79 years.
  2. Cardiovascular Risk Factors, Aging and Dementia (CAIDE) Risk Score ≥6 points.
  3. Cognitive performance at the mean level or slightly lower than expected for age according to local population norms based on the Montreal Cognitive Assessment (MoCA) test and the Consortium to Establish a Registry for Alzheimer's Disease (CERAD) verbal learning test.
  4. Proficiency in the local language (English, Finnish or Swedish)
* Inclusion criteria for metformin/placebo treatment (only for participants in the FINGER 2.0 multimodal lifestyle-based intervention arm)

  1. No diagnosed diabetes or known contraindications to metformin treatment.
  2. Elevated adiposity (BMI≥25 kg/m2 OR waist circumference > 102 cm in men and > 88 cm in women) OR mildly impaired fasting glucose (6.1-6.9 mmol/l).

Exclusion Criteria:

* Main exclusion criteria (all participants)

  1. Dementia or substantial cognitive impairment (e.g., memory clinic referral needed as judged by the study physician).
  2. Current or past use of medications for Alzheimer's Disease or related diseases (e.g., cholinesterase inhibitors, memantine, aducanumab).
  3. Diminished decision-making capacity, not capable of consenting or completing study assessments, based on clinical judgement.
  4. Other known significant neurologic disease (including e.g., Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, brain tumour, progressive, supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma with persistent neurologic sequelae or known structural brain abnormalities).
  5. Any other condition affecting safe engagement in the intervention (e.g., malignant disease, major depression, symptomatic cardiovascular disease, revascularisation within the previous year).
  6. Severe loss of vision, hearing, or communicative ability; conditions preventing cooperation.
  7. Coincident participation in the active phase of another intervention trial.
  8. A member of the household already enrolled in the MET-FINGER trial
* Exclusion criteria for metformin/placebo treatment (only for participants in the FINGER 2.0 multimodal lifestyle-based intervention group)

  1. Use of metformin for any indication.
  2. History of intolerance to metformin used for any indication.
  3. Diabetes diagnosed or suspected at baseline (e.g., HbA1c≥6.5%, fasting glucose ≥7 mmol/l, or 2HPG≥11.1 mmol/l).
  4. Metformin contraindications, e.g., history/presence of known renal or liver disease, congestive heart failure, alcohol abuse, calculated Glomerular Filtration Rate<60 ml/min.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-06-28 (Estimated)

PRIMARY OUTCOMES:
Change in cognition, unit on a scale. | Baseline, 12- and 24-months
  Composite z-score of an extended Neuropsychological Test Battery (NTB) adapted from the FINGER trial and including:
  1. Wechsler Memory Scale Revised (WMS-III, WMS-R) logical memory, immediate
  2. WMS-R logical memory, delayed
  3. WMS-R visual paired associates, immediate
  4. WMS-R visual paired associates, delayed
  5. WMS-R Digit Span, total
  6. Hopkins Verbal Learning Test (HVLT), learning
  7. HVLT, recall
  8. CERAD category fluency
  9. Category fluency (fruits and vegetables)
  10. Trail Making Test (TMT) A
  11. TMT B, shifting score B-A
  12. Stroop Test, shortened 40-stimulus version, condition 2
  13. Stroop Test, condition 3, interference score 3 - 2
  14. Wechsler Adult Intelligence Scale (WAIS) Digit Symbol Substitution Test (DSST).
  The z-score values range from -3 standard deviations to +3 standard deviations of the result distribution with higher score indicating better outcome.

SECONDARY OUTCOMES:
Change in individual cognitive domains, unit on a scale. | Baseline, 12- and 24-months
  Composite z-scores for the:
  * memory
  * executive function
  * processing speed domains that are included in the NTB used as measure for the primary outcome. The z-score values range from -3 standard deviations to +3 standard deviations of the result distribution with higher score indicating better outcome.
Change in functioning level - Clinical Dementia Rating (CDR), unit on a scale | Baseline, 12- and 24-months
  CDR Sum of Boxes (0-18), with lower score indicating a better outcome.
Change in functioning level - Katz index, unit on a scale | Baseline, 12- and 24-months
  Activity of Daily Living, Katz Index. Self-reported questionnaire ranking the independence in six basic daily functions. For each activity, the participant is rated either dependent (0 points) or independent (1 point). The total score ranges 0-6 with a higher score indicating a better outcome.
Change in functioning level - Lawton-Brody scale, unit on a scale | Baseline, 12- and 24-months
  Activity of Daily Living, Lawton-Brody Scale. Self-reported questionnaire assessing the level of functioning in eight daily activities necessary for living in the community. For each activity, the participant is rated either dependent (0 points) or independent (1 point). Score ranges 0-8, with a higher score indicating a better outcome.
Change in healthy lifestyle, unit on a scale. | Baseline, 12- and 24-months
  Healthy Lifestyle Index, a composite score (range 0-24, with higher score indicating a better outcome) including self-reported data on diet, physical activity, smoking and alcohol, and cognitive/social activities.
Change in systolic blood pressure, mmHg. | Baseline, 12- and 24-months
  Lower systolic blood pressure indicates a better outcome.
Change in diastolic blood pressure, mmHg. | Baseline, 12- and 24-months
  Lower diastolic blood pressure indicates a better outcome.
Change in Body Mass Index (BMI), kg/m2. | Baseline, 12- and 24-months
  Calculated using baseline height, with lower BMI value indicating a better outcome.
Change in waist circumference, cm. | Baseline, 12- and 24-months
  Lower value indicates a better outcome, with lower waist circumference value indicating a better outcome.
Change in waist-hip ratio, unit on a scale. | Baseline, 12- and 24-months
  Values ranging up to 1 with lower waist/hip ratio value indicating a better outcome.
Change in blood lipids - Total Cholesterol, mmol/L. | Baseline, 12- and 24-months
  Measured from serum with lower cholesterol value indicating a better outcome.
Change in blood lipids - HDL Cholesterol, mmol/L. | Baseline, 12- and 24-months
  Measured from serum with cholesterol higher value indicating a better outcome.
Change in blood lipids - LDL Cholesterol, mmol/L. | Baseline, 12- and 24-months
  Measured from serum with lower cholesterol value indicating a better outcome.
Change blood triglycerides, mmol/L. | Baseline, 12- and 24-months
  Measured from serum with lower triglycerides value indicating a better outcome.
Change in plasma glucose, mmol/L | Baseline, 12- and 24-months
  Measured from fasting blood sample, with lower glucose value indicating a better outcome.
Change in glycated haemoglobin (HbA1c), % | Baseline, 12- and 24-months
  Measured from fasting blood sample, with lower HbA1c value indicating a better outcome.
Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), unit on a scale. | Baseline, 12- and 24-months
  Calculated using fasting plasma glucose and fasting serum insulin, with lower values indicating a better outcome.
Change in 2-hour plasma glucose, mmol/L. | Baseline, 12- and 24-months
  Measured with Oral Glucose Tolerance Test, only in participants included in the metformin/placebo treatment, and with lower glucose values indicating a better outcome.
Change in dietary intake, unit on a scale. | Baseline, 12- and 24-months
  FINGER Diet Index, with values ranging 0-9, and higher score indicating a better outcome.
Change in physical activity - weekly frequency, unit on a scale. | Baseline, 12- and 24-months
  Self-reported number of sessions moderate-to-vigorous intensity exercise per week. Higher number of sessions indicate a better outcome.
Change in physical activity - Minnesota questionnaire, unit on a scale. | Baseline, 12- and 24-months
  Self-reported physical exercise in the previous two weeks, using a modified version of the Minnesota Leisure Time Physical Activity Questionnaire, as number of sessions and average duration for each of the activities listed in the questionnaire.
  Higher levels of physical activity indicate a better outcome.
Change in physical activity - Actigraph, unit on a scale. | Baseline, 12- and 24-months
  Objective measure of time spent carrying out physical activity using a hip accelerometer (ActiGraph model wGT3X-BT) that the participants will wear for 7 consecutive days.
  Higher levels of physical activity indicate better outcome.
Change in physical functioning - Short Physical Performance Battery (SPPB), unit on a scale. | Baseline, 24-months
  The SPPB is assessed in three domains: balance standing (score range: 0-4), chair standing (score range: 0-4), and gait speed (score range: 0-4). The total score (range: 0-12) is the sum of the three scores. Higher scores indicate a better outcome.
Change in physical functioning - Hand-grip strength, kg | Baseline, 12- and 24-months
  Measured using a hand-grip dynamometer, with higher measures indicating a better outcome.
Change in physical functioning -Timed 10-metre dual task, seconds. | Baseline, 12- and 24-months
  The test measure the time needed to walk 10 metres while carrying out a cognitive task (e.g. naming letters of the alphabet), with shorter times indicating a better outcome.
Change in depressive symptoms, unit on a scale. | Baseline, 12- and 24-months
  Center for Epidemiological Studies Depression scale. Values ranging 0-60, with lower scores indicating a better outcome.
Change in stress-related symptoms, unit on a scale | Baseline, 12- and 24-months
  Perceived Stress Scale. Values ranging 0-40, with lower scores indicating a better outcome.
Change in sleep problems, unit on a scale | 2 years
  Insomnia Severity Index. Values ranging 0-28, with lower scores indicating a better outcome.
Change in health-related quality of life - "Research And Development-36" (RAND-36), unit on a scale | Baseline, 12- and 24-months
  The scale values are ranging 0-100, with higher scores indicating a better outcome.
Change in health-related quality of life - "15D-questionnaire", unit on a scale | Baseline, 12- and 24-months
  The scale values range 0-1, with higher scores indicating a better outcome.
Change in utilisation of health resources, unit on a scale | Baseline, 12- and 24-months
  Number of e.g., hospitalization and doctors appointments, either self-reported and/or, if possible, from General Practitioners, and/or electronic health records of national healthcare registries. Lower use of healthcare resources indicates a better outcome.

OTHER OUTCOMES:
Exploratory - potential interactions between metformin and lifestyle changes | Baseline, 12- and 24-months
  Differences between metformin/placebo treatment groups will be assessed for the lifestyle changes as described for the secondary outcomes.
Exploratory - potential disease-modifying effects - Amyloid β42/40 ratio, unit on a scale | Baseline and 24-months
  Calculated based on blood levels of Amyloid β42 and 40. Possible values range from a minimum of 0, with higher Amyloid β42/40 ratio indicating a better outcome.
Exploratory - potential disease-modifying effects - Neurofilament light chain protein, pg/ml | Baseline and 24-months
  Blood levels of neurofilament light chain protein range from a minimum of 0, with lower levels indicating a better outcome.
Exploratory - potential disease-modifying effects - p-tau 181, ng/ul | Baseline and 24-months
  Blood levels of p-tau 181 range from a minimum of 0, with lower levels indicating a better outcome.
Exploratory - potential disease-modifying effects - p-tau 231, ng/ul | Baseline and 24-months
  Blood levels of p-tau 231 range from a minimum of 0, with lower levels indicating a better outcome.
Exploratory - feasibility of the metformin + lifestyle combination - Adherence to the lifestyle intervention. | 24-months
  Based on consultations and group meetings attended, as well as lifestyle changes implemented. Possible values ranging from a minimum of 0, with higher adherence indicating a better outcome.
Exploratory - feasibility of the metformin + lifestyle combination - Adherence to target metformin dose, unit on a scale | 24-months
  Proportion of participants in each arm of the metformin/placebo treatment who complete the 2-year intervention period on the initially assigned drug dose. Values range 0-1, with higher proportion indicating a better outcome.
Exploratory - feasibility of the metformin + lifestyle combination - Retention rate, unit on a scale | 24-months
  Proportion of randomised participants in each group who complete the 2-year intervention period. Values range 0-1, with higher proportion indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tiia Ngandu, MD, PhD, Principal Investigator — Finnish Institute of Health and Welfare, Finland; Francesca Mangialasche, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (3):
- Finnish Institute of Health and Welfare - THL, Helsinki, Finland
- Karolinska Institutet, Solna, Sweden
- Ageing Epidemiology Research Unit, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The MET-FINGER Steering Committee and Management Group are open to requests from external researchers for data collected in this study. Applicants will be asked to submit a study protocol, including the research question, planned analysis, and data required. Committee will evaluate this plan (i.e., relevance of the research question, suitability of data, quality of proposed analyses, planned/ongoing MET-FINGER analyses, and other matters) on a case-by-case basis and provide the data or reject the request. Shared data will encompass the data dictionary and de-identified data only. Any analysis will be conducted in collaboration with the MET-FINGER Management Group. Access is subject to the MET-FINGER legal framework. An access agreement will be prepared and signed by both parties.
Time Frame: The trial Steering Committee and Management Group will consider applications for data after the trials results have been published and data will be made available according to the terms of the access agreement.
Access Criteria: As described above in the Plan Description.

REFERENCES:
- [Background] Prince M, Ali GC, Guerchet M, Prina AM, Albanese E, Wu YT. Recent global trends in the prevalence and incidence of dementia, and survival with dementia. Alzheimers Res Ther. 2016 Jul 30;8(1):23. doi: 10.1186/s13195-016-0188-8. PMID 27473681
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Kivipelto M, Mangialasche F, Snyder HM, Allegri R, Andrieu S, Arai H, Baker L, Belleville S, Brodaty H, Brucki SM, Calandri I, Caramelli P, Chen C, Chertkow H, Chew E, Choi SH, Chowdhary N, Crivelli L, Torre R, Du Y, Dua T, Espeland M, Feldman HH, Hartmanis M, Hartmann T, Heffernan M, Henry CJ, Hong CH, Hakansson K, Iwatsubo T, Jeong JH, Jimenez-Maggiora G, Koo EH, Launer LJ, Lehtisalo J, Lopera F, Martinez-Lage P, Martins R, Middleton L, Molinuevo JL, Montero-Odasso M, Moon SY, Morales-Perez K, Nitrini R, Nygaard HB, Park YK, Peltonen M, Qiu C, Quiroz YT, Raman R, Rao N, Ravindranath V, Rosenberg A, Sakurai T, Salinas RM, Scheltens P, Sevlever G, Soininen H, Sosa AL, Suemoto CK, Tainta-Cuezva M, Velilla L, Wang Y, Whitmer R, Xu X, Bain LJ, Solomon A, Ngandu T, Carrillo MC. World-Wide FINGERS Network: A global approach to risk reduction and prevention of dementia. Alzheimers Dement. 2020 Jul;16(7):1078-1094. doi: 10.1002/alz.12123. Epub 2020 Jul 5. PMID 32627328
- [Derived] Barbera M, Lehtisalo J, Perera D, Aspo M, Cross M, De Jager Loots CA, Falaschetti E, Friel N, Luchsinger JA, Gavelin HM, Peltonen M, Price G, Neely AS, Thunborg C, Tuomilehto J, Mangialasche F, Middleton L, Ngandu T, Solomon A, Kivipelto M; MET-FINGER study team. A multimodal precision-prevention approach combining lifestyle intervention with metformin repurposing to prevent cognitive impairment and disability: the MET-FINGER randomised controlled trial protocol. Alzheimers Res Ther. 2024 Jan 31;16(1):23. doi: 10.1186/s13195-023-01355-x. PMID 38297399